CLINICAL TRIAL: NCT06027853
Title: Clinical Study to Evaluate the Safety and Efficacy of iPSC NK Cells Targeting CLL1 in Patients With Relapsed/Refractory AML
Brief Title: Natural Killer(NK) Cell Therapy Targeting CLL1 in Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Qihangene Biotech Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, He Huang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH-CLL1-01
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-NK cell therapy in Adult subjects with r/r AML (Experimental): CAR-NK cell therapy in Adult subjects with r/r AML
  Interventions: Drug: CLL1 CAR-NK cell injection

INTERVENTIONS:
Drug: CLL1 CAR-NK cell injection — Drug: CLL1 NK cell therapy Drug: Cyclophosphamid Lympho-conditioning Agent Drug: Fludarabine Lympho-conditioning Agent
  Drug: VP-16 Lympho-conditioning Agent

SUMMARY:
This is a phase 1, first-in-human (FIH), open-label, multicohort study to evaluate the safety, tolerability and preliminary efficacy of CLL1 target CAR iPSC NK cells in patients with relapsed/refractory AML

DETAILED DESCRIPTION:
Acute myelogenous leukemia (AML) is a potentially cur-able disease; 70% of newly diagnosed patients achievecomplete remission with first-line therapy, but prognosisworsens for relapsed disease in both pediatric and adultpatients. CLL-1 has attracted the researchers' attention due to its high expression in AML while being absent in normal hematopoietic stem cell. Accumulating evidence have demonstrated CLL-1 is an ideal target for AML.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old.
2. Confirmed diagnosis of r/r AML
3. CLL1 expression is positive in AML blasts.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤1 and life expectancy greater than 12 weeks.
5. Adequate organ and marrow function, as defined below:

   1. Blood creatinine (Cr) ≤ 2 x ULN or calculated creatinine clearance (Cockcroft- Gault formula) ≥ 50 mL/min;
   2. Total bilirubin (TBIL) ≤ 2 x the ULN;
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN;
   4. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
6. Females of childbearing potential must have a negative serum pregnancy test.
7. Donor specific antibody (DSA) is negative: MFI <= 2000.
8. Provision of signed and dated informed consent form (ICF).

Exclusion Criteria:

1. Allergic to drug used in this study.
2. Subjects received any antitumor therapy as follows, prior to first NK infusion:

   1. Systemic steroid therapy within 3 days (except physiological replacement therapy);
   2. Systemic antitumor therapy within 2 weeks or at least 5 half-lives, whichever is less;
   3. Radiotherapy within 4 weeks;
   4. Donor lymphocyte infusion within 6 weeks;
   5. Intrathecal treatment within 1 week;
   6. CAR-T therapy, CAR-NK therapy, or any other genetically modified cell therapy product within 6 months;
3. History of allogeneic stem cell transplantation.
4. Received the vaccine within 4 weeks prior to the first infusion and/or expected to require vaccination from the study period to 12 weeks after the last infusion.
5. Active central nervous system Leukemia.
6. Acute Promyelocytic Leukemia (APL).
7. History of other malignant tumors, except for those who have achieved complete remission more than 5 years after radical treatment without any signs of recurrence.
8. Active autoimmune diseases.
9. History of central nervous system disease or meningeal involvement such as epilepsy, paralysis, aphasia, stroke, etc.
10. Serious cardiovascular and cerebrovascular diseases:

    1. Severe heart rhythm or conduction abnormalities, corrected QT interval (QTc)≥480 ms;
    2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events within 6 months prior to first infusion;
    3. New York Heart Association (NYHA) class II or above congestive heart failure or left ventricular ejection fraction (LVEF) <50% in color Doppler echocardiography;
    4. Hypertension that cannot be controlled by drug.
11. Active pulmonary infection; SpO2 ≤90%; Pulmonary embolism, chronic obstructive pulmonary disease, or interstitial lung disease.
12. Uncontrolled bacterial, fungal, or viral infection. Known HIV infection, active Hepatitis B (HBV) or Hepatitis C (HCV) infection.
13. History of substance abuse.
14. Toxicity induced by previous therapy not recovered to ≤ grade 2(NCI-CTCAE v5.0).
15. Large surgical treatment within 4 weeks prior to first infusion, not including diagnostic biopsy.
16. Pregnant/breastfeeding women.
17. Investigator-assessed presence of any medical or social issues that are likely to interfere with study conduct or may cause increased risk to subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 Days from first dose of iPSC NK cell infusion
  Safety and Tolerability
Incidence of subjects with Dose Limiting Toxicities within each dose level cohort | 28 Days from first dose of iPSC NK cell infusion
  Tolerability

SECONDARY OUTCOMES:
Determination of the pharmacokinetics (PK) of iPSC NK cells in peripheral blood | Up to approximately 2 years after last dose of iPSC NK cell infusion
  The PK of iPSC NK in peripheral blood will be reported as the relative percentage of product DNA versus patient DNA (% chimerism) measured from blood samples at the specified time points

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- Clinical research ethics committee of the first affiliated hospital, college of medicine, zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No